CLINICAL TRIAL: NCT06355531
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Assess the Efficacy, Safety, and Pharmacokinetics of FNP-223 (Oral Formulation) to Slow the Disease Progression of Progressive Supranuclear Palsy (PSP) (PROSPER)
Brief Title: A Study to Assess the Efficacy, Safety, and Pharmacokinetics of FNP-223 to Slow Progression of Progressive Supranuclear Palsy (PSP)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNP223-CT-2301
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy; Disease progression; FNP-223
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Disease Progression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FNP-223 (Experimental): Participants will receive FNP-223 orally (PO), 3 times daily (TID).
  Interventions: Drug: FNP-223
- Placebo (Placebo Comparator): Participants will receive matching placebo, PO, TID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FNP-223 — Oral tablets
  Arms: FNP-223
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
PROSPER trial is a trial to assess the efficacy of FNP-223 in slowing disease progression in participants with PSP as measured by the PSP Rating Scale (PSPRS) over 52 weeks and to assess the safety and tolerability of FNP-223 for 52 weeks in participants with PSP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 50 to 80 years, inclusive, at the time of informed consent.
* Diagnosis of possible or probable PSP of the Richardson's Syndrome (PSP-RS) phenotypes according to the Movement Disorders Society's Progressive Supranuclear Palsy (MDS PSP) clinical features criteria. At least 1 (either 1 or both) of the following 2 items must be met:

  1. Vertical supranuclear gaze palsy.
  2. Slowing of vertical saccades AND postural instability with falls within the first 3 years of PSP symptoms.
* Presence of PSP symptoms within ≤3 years prior to screening.
* MoCA score ≥23
* Full 28-item PSPRS score ≤40.
* Able to ambulate independently or with minimal assistance defined as the ability to take at least 10 steps (stabilization of 1 arm [ie, use of cane]).
* Body weight range ≥43 kg/95 lbs to ≤120 kg/265 lbs.
* Reside outside a skilled nursing facility or dementia care facility, except for participants residing in an assisted living facility.
* Has a caregiver or study partner who will accompany them to the study visits. The caregiver or study partner must be a person who has frequent contact (at least 7 hours per week at 1 time or in different days) with the participant and is able to provide information about the participant's medication and overall condition. Prior to the conduct of any study procedures, the caregiver or study partner must be willing to sign the independent ethics committee (IEC)/institutional review board (IRB) approved informed consent.

Exclusion Criteria:

Non-PSP- RS Movement Disorders or other central nervous system (CNS) Diseases

* Score of 3 on any functional domain in the PSP-CDS.
* Participants with known PSP genetic mutation (based on familiar or clinical history).
* Evidence of other neurological disorder that could explain signs of PSP (eg, Parkinson's disease, Alzheimer disease, etc.).
* Brain magnetic resonance imaging (MRI) within 1 year of screening consistent with:
* Primary degenerative diseases other than PSP.

Procedures

* For the optional substudy only: Contraindication or refusal to undergo 2 lumbar punctures for obtaining CSF.
* Contraindication or inability to tolerate MRI for screening MRI and volumetric brain MRI assessments throughout the substudy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 52 in the PSPRS Outcome | Baseline to Week 52
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Baseline to Week 52
  Clinically significant changes in vital signs, clinical laboratory evaluations, physical examinations, and electrocardiogram (ECG) are included in TEAEs.
Number of Participants Experiencing Serious Adverse Events (SAEs) | Baseline to Week 52

SECONDARY OUTCOMES:
Change From Baseline to Week 52 in Clinical Global Impression of Severity Scale (CGI-S) | Baseline to Week 52
Change From Baseline to Week 52 Participant Global Impression of Severity Scale (PGI-S) | Baseline to Week 52
Change From Baseline to Week 52 in Caregiver Global Impression of Severity Scale (CaGI-S) | Baseline to Week 52
Slope of Decline in PSPRS | Baseline to Week 52
Change From Baseline to Week 52 in Individual Subitems of PSPRS | Baseline to Week 52
Change From Baseline to Week 52 in Schwab and England Activities of Daily Living Scale | Baseline to Week 52
Change From Baseline to Week 52 in PSP Clinical Deficits Scale (PSP-CDS) | Baseline to Week 52
Change From Baseline to Week 52 in Montreal Cognitive Assessment (MoCA) | Baseline to Week 52
Change From Baseline to Week 52 in PSP Quality of Life Scale (PSP-QoL) | Baseline to Week 52
Pharmacokinetic characterization of FNP-223 | At Week 4 and Week 16
  Mean plasma concentration of FNP-223.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (12):
  - The Neurology Center of Southern California - Carlsbad, Carlsbad, California
  - UCSF Weill Institute for Neurosciences, San Francisco, California
  - Rocky Mountain Movement Disorders Center, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Augusta University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Robert & John M. Bendheim Parkinson and Movement Disorders Center at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Duke Neurology, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Central Texas Neurology Consultants, Round Rock, Texas
- France (5):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital de la Timone, Marseille
  - L'Hôpital Universitaire Carémeau, Nîmes
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - Hôpital Pierre-Paul Riquet, Toulouse
- Germany (4):
  - Neurologisches Fachkrankenhaus für Bewegungsstörungen/Parkinson, Beelitz
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Leipzig, Leipzig
  - Ludwig-Maximilians-Universität München (LMU), Munich
- Pécsi Tudományegyetem Általános Orvostudományi Kar, Pécs, Hungary
- Italy (5):
  - IRCCS Istituto Delle Scienze Neurologiche di Bologna, Bologna
  - Azienda Ospedale Università di Padova, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - San Raffaele Pisana, Roma
  - Azienda Ospedaliera Universitaria San Giovanni di Dio Ruggi d'Aragona, Salerno
- Poland (2):
  - Neurologia Śląska Centrum Medyczne, Katowice
  - Mazowiecki Szpital Bródnowski w Warszawie, Warsaw
- Portugal (2):
  - Hospital de Braga, Braga
  - Campus Neurológico Senior - Torres Vedras, Torres Vedras
- Spain (9):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (4):
  - University of Cambridge, Cambridge
  - University College London Hospitals, London
  - Newcastle Upon Tyne Hospitals, Newcastle
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pokorny R, Ryan JM, Abd-Elaziz K, van den Berg F, Rabiner E, Searle GE, Schneider M, Wiessner C, Stallaert JF, Permanne B, Quattropani A, Beher D. Safety, Tolerability, Pharmacokinetics, and Brain Target Occupancy of the OGA Inhibitor ASN90 in Healthy Participants. Mov Disord. 2025 Nov 15. doi: 10.1002/mds.70104. Online ahead of print. PMID 41239890